CLINICAL TRIAL: NCT02454920
Title: Measurement of the Distance Between the Limbus and Insertion of Extraocular Muscles Using Anterior Segment Optical Coherence Tomography
Brief Title: Measurement of Insertion of Extraocular Muscles Using Anterior Segment Optical Coherence Tomography
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hilda Capo, Professor of Clinical, University of Miami
Other Study IDs: 20150332
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Strabismus; Tomography, Optical Coherence
Keywords: Strabismus; Optical Coherence Tomography; Extraocular muscles
MeSH Terms: conditions — Strabismus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Study designed to determine the ability and accuracy of anterior segment optical coherence tomography (AS-OCT) to measure the distance between the corneoscleral limbus and the insertion site of the extraocular muscles (EOM) in adults with and without previous strabismus surgery. And to compare in surgical patients the pre-operative AS-OCT limbal-muscle insertion distance measurement to the intraoperative limbal-muscle insertion measurement using calipers (gold standard).

DETAILED DESCRIPTION:
The treatment of strabismus is often surgical. A better surgical plan would be possible if the exact limbus-insertion distance of the extraocular muscles was known. The clinical ophthalmologic examination, such as slit lamp biomicroscopy, cannot elucidate the muscle insertion position prior to surgery. This information is especially important in patients who have undergone prior strabismus surgery. In these patients, previous surgical data may not be available or the muscle insertion may be in a different location than expected. Thus, a preoperative imaging study that could accurately locate the muscle insertion may be useful for designing the surgical plan, possibly improving the success of the surgery, and reducing operative time and intraoperative complications.

Previous studies that used computed tomography (CT) scans and high-resolution magnetic resonance imaging (MRI), have failed to reliably detect the rectus muscle insertions. Ocular ultrasound allows anatomic visualization of the EOM, but has a low image resolution. Ultrasound biomicroscopy (UBM), can accurately measure the limbus-insertion distance, however, it induces significant measurement errors due to the pressure applied to the globe during examination. The recent advances in AS-OCT imaging allow non-invasive, detailed, cross-sectional examination of anterior segment structures by generating a two-dimensional high resolution image from a reflected light beam. Two previous studies have successfully used AS-OCT to analyze EOM insertions, but the number of participants was small and patients with previous strabismus muscle surgery were not included.

The investigators purpose is to gather limbus-EOM insertion distance data using the AS-OCT in a greater number of patients, include patients who have undergone previous strabismus procedures, and correlate AS-OCT measurements with intraoperative findings in those patients undergoing strabismus surgery.

Procedures

1. After recruitment, a written consent will be obtained from subjects who agree to participate.
2. A review of medical records will be performed to obtain demographics data, type of strabismus, history of previous eye surgery, etc (see Data Collection Sheet)
3. AS-OCT imaging of the rectus muscles will be performed in all patients using the Visante (Visante AS-OCT; Carl Zeiss Meditec) and/or Heidelberg Spectralis (Spectralis AS-OCT; Heidelberg Engineering) instruments.
4. For patients undergoing strabismus surgery, the distance from the corneoscleral limbus to the insertion site of the rectus muscles will be measured with calipers at the time of the surgery.
5. After the surgery, AS-OCT imaging of the rectus muscles will be performed during routinely scheduled post-operative clinic visits.

All acquired images will be stored in the Bascom Palmer Eye Institute MERGE HealthCare Completes Acquisition of Ophthalmic Imaging Systems (OIS), a clinical imaging storage system, which is secured against unauthorized access. All background information will be entered into REDCAP data capturing system by one of the investigators and be accessible only to the investigators (http://www.project-redcap.org/).

The AS-OCT devices that will be used are commercially available, FDA approved, and routinely used in clinical settings to evaluate the anterior and posterior segments of the eye. There are no experimental imaging procedures planned for the purpose of this study. All imaging acquisition protocols have been well-established and are non-invasive. There is no contact with the eye during image acquisition. This exposes the subjects to no greater than minimal risk as the result of participating in this study.

All eligible adult patients who are undergoing strabismus evaluation at the Bascom Palmer Eye Institute will be invited to participate. The consent processes will occur during the clinic visit. The study does not involve any additional clinic visits. The patient will have ample opportunity to discuss the study, review the consent form, and sign the consent form during the course of the visit. This study will follow the SOP: Informed Consent Process for Research (HRP-090).

Non-English Speaking Subjects We will exclude patients whose English proficiency precludes reading the form and understanding its contents.

ELIGIBILITY:
Inclusion Criteria:

* All patients age ≥ 18 years undergoing a strabismus evaluation at the Bascom Palmer Eye Institute will be invited to participate. Members of the study team will be involved in the clinical evaluation. The physician will determine if the patient has strabismus and whether strabismus surgery is advisable.

Exclusion Criteria:

1. Patient who is unwilling to participate the study.
2. A clinical scenario in which AS-OCT examination is not likely to be successful (e.g. an uncooperative patient).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients age greater then 18 years undergoing a strabismus evaluation at the Bascom Palmer Eye Institute
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Limbus to extraocular muscles insertion distance | Baseline measurement
  Measurement of the limbus to insertion distance with OCT

SECONDARY OUTCOMES:
Comparison between intra operative and OCT measurements of the distance from the limbus to extraocular muscles insertion | From date of baseline to date of surgery
  Measurement of the limbus to insertion distance with OCT (mm) and measurement of the limbus to insertion distance with a caliper at time of surgery (mm)

CONTACTS AND LOCATIONS:
Overall Officials: Hilda Capo, MD, Principal Investigator — Professor

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liu X, Wang F, Xiao Y, Ye X, Hou L. Measurement of the limbus-insertion distance in adult strabismus patients with anterior segment optical coherence tomography. Invest Ophthalmol Vis Sci. 2011 Oct 28;52(11):8370-3. doi: 10.1167/iovs.11-7752. PMID 21948556
- [Background] Park KA, Lee JY, Oh SY. Reproducibility of horizontal extraocular muscle insertion distance in anterior segment optical coherence tomography and the effect of head position. J AAPOS. 2014 Feb;18(1):15-20. doi: 10.1016/j.jaapos.2013.11.005. PMID 24568976
- [Background] Dai S, Kraft SP, Smith DR, Buncic JR. Ultrasound biomicroscopy in strabismus reoperations. J AAPOS. 2006 Jun;10(3):202-5. doi: 10.1016/j.jaapos.2006.01.209. PMID 16814170